CLINICAL TRIAL: NCT06747065
Title: Retrospective International Multicenter Study Comparing Polyurethan Versus Non-polyurethan Covered Implants in Immediate Prepectoral Implant-based Breast Reconstruction in the Setting of Postmastectomy Radiotherapy: the PRExRT Study
Brief Title: Polyurethan Versus Non-polyurethan Covered Implants in Combination With Radiotherapy
Acronym: PRExRT
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-02438; bb24weber3
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Mastectomy; Lymphedema; Breast Cancer
Keywords: immediate implant-based breast reconstruction (IBBR); postmastectomy radiotherapy (PMRT); Polyurethan covered implant
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PU covered implants: prepectoral IBBR with a PU covered implant followed by radiotherapy
  Interventions: Procedure: Radiotherapy
- non-PU covered implants: prepectoral IBBR with a non-PU covered implant followed by radiotherapy
  Interventions: Procedure: Radiotherapy

INTERVENTIONS:
Procedure: Radiotherapy — Radiotherapy post-mastectomy prepectoral implant-based breast reconstruction (IBBR)

SUMMARY:
The purpose of this multicenter retrospective cohort study is to determine the effect of radiotherapy on capsular contraction and implant loss rates in patients undergoing prepectoral immediate implant-based breast reconstruction (IBBR) comparing Polyurethan (PU) and non-PU covered implants.

DETAILED DESCRIPTION:
Breast cancer affects 2.6 million women worldwide annually, with surgery as the standard treatment for 95% of cases. Rising mastectomy rates, due to advanced diagnostic tools and patient preferences, make immediate breast reconstruction crucial for improving quality of life for around 650,000 women each year. Prepectoral implant-based breast reconstruction (IBBR) has become a preferred approach due to advancements like synthetic meshes, acellular dermal matrices (ADM), and polyurethane (PU) covered implants, which show promise in reducing complications such as capsular contracture, implant loss, and breast animation deformities. Radiotherapy (RT), however, increases these risks, especially for capsular contracture, underscoring the need for strategies to mitigate such outcomes.

This multicenter retrospective cohort study will investigate the impact of radiotherapy on complications such as capsular contracture and implant loss in patients with breast cancer who underwent mastectomy and prepectoral IBBR. The study will compare outcomes between PU and non-PU covered implants using data from approximately 30 international sites. Patient information will be extracted from hospital records, coded for confidentiality, and analyzed statistically to achieve the study's objectives of improving post-reconstruction outcomes and quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with signed General consent or study specific consent form
* Patients with confirmed diagnosis of primary or recurrent breast cancer
* Patients undergoing nipple - or skin-sparing mastectomy with prepectoral IBBR (all types of implants, with or without mesh, all types of biologic and synthetic mesh, one- or two- stage) in the setting of PMRT (or any type or RT before reconstruction) between 2016 and 2022.
* Patients undergoing two-stage IBBR with radiotherapy to the expander before reconstruction with implant.
* Patients with recurrent breast cancer after breast conserving surgery and radiotherapy.
* Follow up must be at least 2 years after IBBR.
* Patients aged 18 and above will be eligible for inclusion.

Exclusion Criteria:

* Patients who have explicitly refused the further use of their data through a consent declaration.
* Patients undergoing subpectoral IBBR or autologous reconstruction as initial type of reconstruction.
* No radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: data will be collected from patient hospital records, including approximately 30 international sites
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
capsular contracture | 2-6 years post-surgery
  capsular contracture rate in women with IBBR in combination with RT comparing the use of PU with non-PU implants

SECONDARY OUTCOMES:
implant loss rate | 2-6 years post-surgery
  To determine the implant loss rate in women with IBBR in combination with RT comparing the use of PU with non-PU implants
re-surgery rate | 2-6 years post-surgery
  To determine the re-surgery rate in women with IBBR in combination with RT comparing the use of PU with non-PU implants
hematoma rate | 2-6 years post-surgery
  To determine the hematoma rate in women with IBBR in combination with RT comparing the use of PU with non-PU implants
infection rate | 2-6 years post-surgery
  To determine the infection rate in women with IBBR in combination with RT comparing the use of PU with non-PU implants
implant exchange rate | 2-6 years post-surgery
  To determine the implant exchange rate in women with IBBR in combination with RT comparing the use of PU with non-PU implants

CONTACTS AND LOCATIONS:
Overall Officials: Walter Weber, Prof. Dr., Principal Investigator — Universitätsspital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland